CLINICAL TRIAL: NCT04864795
Title: Cardiovascular and Renal Treatment in Heart Failure Patients With Hyperkalaemia or at High Risk of Hyperkalaemia (CARE-HK in HF Registry)
Brief Title: Cardiovascular and Renal Treatment in Heart Failure Patients With Hyperkalaemia or at High Risk of Hyperkalaemia
Acronym: CARE-HK
Status: Completed | Type: Observational
Sponsor: Vifor (International) Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Other Study IDs: HQ-NIS-CHF-07.2020
Record Dates: First submitted 2021-04-06; First posted 2021-04-29 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure; Hyperkalemia
MeSH Terms: conditions — Heart Failure; Hyperkalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single Cohort: Patient data will be collected from patient records and/or during a routine clinical visit. This will include treatments prescribed, routine assessments and measurements collected at routine clinical visits, as well as hospitalisations and other relevant patient data.

SUMMARY:
The CARE-HK in HF is a registry study based on the hypothesis that adherence to guidelines is associated with improved real-world outcomes for heart failure (HF) patients. For the purpose of this study, adherence to guidelines is defined as adherence to RAASi treatment recommendations, according to the AHA/ACC and ESC guidelines. Objectives relating to patiromer effectiveness will only be evaluated if a sufficient number of patients are available.

The study aims to evaluate in patients at high risk of hyperkalaemia; patients treated with ACEi/ARB/ARNi, and either treated with or candidates for treatment with MRA.

DETAILED DESCRIPTION:
The study will have an enrolment period of approximately 24 months, and each patient will be followed prospectively for at least 6 months. Each patient is expected to contribute to the study data collection until study end or until premature discontinuation, whichever occurs first (i.e., due to death, withdrawal of consent, or lost to follow-up).

At enrolment (informed consent signed by patient), relevant patient data will be retrospectively extracted from medical records for the 24 months prior to enrolment or since the time of HF diagnosis.

There are no visits or procedures associated with the study, patients will follow routine clinical care, which may include in-person and/or virtual visits. The study protocol does not recommend the use of any specific treatments and no study medication is provided as part of participation. The nature and heterogeneity of HF means patients will be treated with different treatments over the course of the study, and at the discretion of their treating physician.

Patient data will be collected from patient records and/or during a routine clinical visit and will be entered into the electronic Case Report Form (eCRF) via an electronic data capture (EDC) system. This will include treatments prescribed, routine assessments and measurements (e.g., laboratory parameters) collected at routine clinical visits, as well as hospitalisations and other relevant patient data. Protocol version 3.0, 19-Jul-2023

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged ≥18 years at enrolment.
2. Patient diagnosed with chronic HF ≥3 months prior to signature of informed consent.
3. Patient has at least 1 record of LVEF documented in patient medical record in the 24 months prior to signature of informed consent. NOTE: If the proportion of patients with HFpEF exceeds 20% of the target sample size, enrolment of patients with an LVEF ≥50% may be capped.
4. Patient treated with ACEi/ARB/ARNi at enrolment.
5. Patient treated with or a candidate for treatment with MRA per a relevant treatment guideline (e.g., HF, CKD, resistant hypertension) at enrolment.
6. Patient at increased risk of hyperkalaemia due to one or more of the following:

   1. Current hyperkalaemia (sK+ >5.0 mEq/l) at enrolment
   2. Record of documented hyperkalaemia (sK+ >5.0 mEq/l) in the 24 months prior to signature of informed consent
   3. eGFR <45 ml/min/1.73 m2, or CKD Stage ≥3b.
7. Patient judged by the Investigator to have sufficient cognitive ability to participate.
8. Signed informed consent provided

Exclusion Criteria:

1. Patient on renal replacement therapy or mechanical circulatory support.
2. Disease other than HF with expected survival <1 year.
3. Patient is participating in, or being screened for, an interventional trial, with the exception of interventional trials relating to SARS-CoV-2.
4. Patient already found to be intolerant to MRA for reasons other than hyperkalaemia or renal impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To the extent possible, representative sites (e.g., cardiologists and nephrologists) reflective of the treatment patterns within each country will be recruited. All patients treated for chronic HF during the enrolment period will be assessed for eligibility, and all eligible patients will be consecutively proposed to enrol in the study as they present for a routine clinical visit (in-person or virtual visits) in order to avoid potential selection bias.
Sampling Method: Non-Probability Sample
Enrollment: 2636 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients by RAASi optimisation | at 6-months intervals
  overall
Percentage of patients by RAASi dose modification following hyperkalaemic episodes | at 6-month intervals after a hyperkalaemic episode
  RAASi
Comparison of percentage of patients with RAASi treatment optimisation between patiromer treated and untreated patients following hyperkalaemic | at 6-months following enrolment
  episodes

SECONDARY OUTCOMES:
Occurrence and incidence of hyperkalaemia events by RAASi treatment optimisation | at 6-months following enrolment
  RAASi
Description of physician provided reasons for treatment decisions at initiation or modification/discontinuation of RAASi treatment | up to 6 months following enrolment
  RAASi
Description and change of disease status measured by patient reported outcome (PRO) by RAASi treatment optimisation | at enrolment and at approximately 6-months intervals
  Kansas City Cardiomyopathy Questionnaire (KCCQ)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Wächter, Study Chair — Vifor International
Locations (116):
- United States (52):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UC San Diego Sulpizio Cardiovascular Center, La Jolla, California
  - Amicis Research Center, Northridge, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Bethesda Hospital East, Boynton Beach, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Inpatient Research Clinic, LLC, Hialeah, Florida
  - Clearwater Cardiovascular Consultants, Largo, Florida
  - D&H National Research Centers, Miami, Florida
  - Southwest Florida Research, LLC, Naples, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - Clearwater Cardiovascular and Interventional Consultants, Safety Harbor, Florida
  - Florida Cardiology P.A, Winter Park, Florida
  - IACT Health, Columbus, Georgia
  - Cardiology Care Clinics, Eatonton, Georgia
  - NSC Research, Johns Creek, Georgia
  - Chicago Medical Research, LLC, Hazel Crest, Illinois
  - Prairie Cardiovascular Consultants, Ltd., Springfield, Illinois
  - Cardiovascular Medicine, P.C., Davenport, Iowa
  - Central Cardiology Associates, Elizabethtown, Kentucky
  - Maine Health, Biddeford, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - TidalHealth Peninsula Regional Inc., Salisbury, Maryland
  - Ascension St. Mary's Hospital, Saginaw, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - St. Louis Heart and Vascular, Bridgeton, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - St. Louis University, St Louis, Missouri
  - Logan Health Research, Kalispell, Montana
  - Virtua Medical Group PA, Marlton, New Jersey
  - Raritan Bay Primary and Cardiology Associates, Matawan, New Jersey
  - The Heart House, Sewell, New Jersey
  - Albany Stratton VA Medical Center, Albany, New York
  - Capital Cardiology Associates, Albany, New York
  - South Shore University Hospital, Bay Shore, New York
  - Focus Clinical Research Solutions, Charlotte, North Carolina
  - Nephrology Associates of Greater Cincinnati, Cincinnati, Ohio
  - Rama Research LLC, Marion, Ohio
  - The Heart and Medical Center, Durant, Oklahoma
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - East Texas Cardiology PA, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Texas Cardiology Associates of Houston, Kingwood, Texas
  - Complete Heart Care, McKinney, Texas
  - Baylor Scott & White Round Rock, Round Rock, Texas
  - Baylor Scott & White Health - Temple, Temple, Texas
  - Victoria Heart & Vascular Center, Victoria, Texas
  - Richmond Cardiology Associates, Mechanicsville, Virginia
  - William S. Middleton Memorial VA Hospital, Madison, Wisconsin
- Austria (6):
  - KH St. Josef Braunau, Braunau am Inn
  - LKH Universitatklinikum Graz, Graz
  - Ordensklinkum Linz Elisabethinen, Linz
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
  - Imed-19 privat, Vienna
  - Klinik Floridsdorf, Vienna
- Belgium (6):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - AZ Sint-Blasius, Dendermonde
  - CHU de Liège, Liège
  - AZ Glorieux, Ronse
- Italy (12):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna, Ferrara
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, Foggia
  - A.O.U. Policlinico di Modena, Modena
  - Centro Cardiologico Monzino-IRCCS, Monza
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Arcispedale S. Maria Nuova Azienda Ospedaliera di Reggio Emilia, Reggio Emilia
  - IRCCS San Raffaele Pisana, Roma
  - IRCCS Ospedale Policlinico San Martino, San Martino
  - Azienda Servizi Sanitari 1 Triestina, Trieste
- Spain (23):
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Juan Ramon Jimenez Hospital, Huelva
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Puerto Real, Puerto Real
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hosp. Universitari Sant Joan de Reus, Tarragona
- Switzerland (6):
  - Kantonsspital Aarau AG, Aarau
  - University Hospital Basel, Basel
  - Hôpitaux Universitaires de Genève - HUG, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
- United Kingdom (11):
  - Buckinghamshire Healthcare NHS Trust, Amersham
  - Bradford Royal Infirmary, Bradford
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Northwick Park Hospital, Harrow
  - Royal Liverpool University Hospital, Liverpool
  - Barts Health NHS Trust, London
  - King's College Hospital, London
  - William Harvey Clinical Research Centre, London
  - Royal Victoria Infirmary, Newcastle
  - Derriford Hospital, Plymouth
  - Whiston Hospital, Rainhill

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be requested 6 months after the primary publication for the entire prospective observation period.
  Data will be available 5 years for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and the study sponsor and researchers must sign a data sharing agreement.

REFERENCES:
- [Derived] Greene SJ, Sauer AJ, Bohm M, Bozkurt B, Butler J, Cleland JGF, Coats AJS, Desai NR, Grobbee DE, Kelepouris E, Pinto F, Rosano G, Donachie V, Fabien S, Waechter S, Crespo-Leiro MG, Hulsmann M, Kempf T, Pfister O, Pouleur AC, Saxena M, Schulz M, Volterrani M, Anker SD, Kosiborod MN. Management of patients with heart failure at high risk of hyperkalaemia: The CARE-HK in HF registry. Eur J Heart Fail. 2025 Nov;27(11):2410-2421. doi: 10.1002/ejhf.3800. Epub 2025 Aug 11. PMID 40788620